CLINICAL TRIAL: NCT06653192
Title: Endoscopic Ultrasound-Guided Biliary Drainage With Lumen-Apposing Stent vs Classical ERCP for First-line Therapy of Malignant Distal Biliary Obstruction: An Open-label, Multicenter Randomized Trial (CARPEDIEM Trial)
Brief Title: EUS-guided Choledochoduodenostomy vs ERCP as First Line in Malignant Distal Obstruction (CARPEDIEM Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Hospital Clínico Universitario de Valencia (Other); Hospital General Universitario de Alicante (Other); Hospital General Universitario de Castellón (Other); Complejo Hospitalario Universitario de Santiago (Other); University Hospital Virgen de las Nieves (Other); Complejo Hospitalario de Navarra (Other); Hospital de Sant Pau (Other); University of Salamanca (Other)
Responsible Party: Principal Investigator, Joan B Gornals, PhD and Head of Interventional Endoscopy Unit, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARPEDIEM
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Malignant Biliary Obstruction; Pancreatic Cancer; Biliary Tract Neoplasms
Keywords: Choledochoduodenostomy; Therapeutic endoscopy; Biliary Drainage; Lumen apposing metal stent; ERCP; Biliopancreatic malignancy
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ERCP with SEMS (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) with deployment of a self-expandable metallic stent (SEMS). Gold standard in malignant distal biliary obstruction (MDBO) in current practice.
  ERCP technique: Cannulation with papillotome (advanced cannulation techniques are allowed). Sphincterotomy. Self-expandable metallic stent (SEMS) deployment.
  Interventions: Procedure: Endoscopic biliary drainage; Device: Self-expandable metallic stent (SEMS)
- EUS-CDS with LAMS-Pigtail (Experimental): Echoendoscopy-guided Choledochoduodenostomy (EUS-CDS) with deployment of a lumen-apposing metal stent (LAMS) and axis-orienting double-pigtail plastic stent throug LAMS.
  EUS-CDS technique: Diagnostic EUS. Classic or free-hand with preloaded guidewire choledochoduodenostomy with LAMS. Pneumatic dilation whithin LAMS is allowed. In case of bile duct < 15mm is mandatory the 'push' technique. Deployment of a pigtail coaxial to LAMS.
  Interventions: Procedure: Endoscopic biliary drainage; Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS)

INTERVENTIONS:
Procedure: Endoscopic biliary drainage — Decompression of the bile duct by endoscopic aproach.
Device: Self-expandable metallic stent (SEMS) — Self-expandable metallic stent (SEMS) deployment:
  Covering: Uncovered or Partially Covered. Non covered if gallbladder is present.
  Size: 10x40mm or 10x60mm or 10x80mm.
  Arms: ERCP with SEMS
Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS) — Lumen-apposing metal stent (LAMS) with coaxial double-pigtail plastic stent (DPPS) deployment:
  LAMS size: 6x8mm or 8x8mm. Consider 10x10mm if bile duct > 18mm. DPPS size: 7Fr x 3-7cm.
  Arms: EUS-CDS with LAMS-Pigtail

SUMMARY:
The aim of this clinical trial is to evaluate the biliary drainage technical failure rate and/or the postprocedure acute pancreatitis rate between EUS-CDS vs ERCP procedures in patients with distal malignant biliary obstruction.

DETAILED DESCRIPTION:
Ecoendoscopy-guided choledochoduodenostomy (EUS-CDS) has been extended as a second line treatment in cases of ERCP failure in malignant distal biliary obstruction (MDBO). However, there are clinical trials which have compared it with ERCP as a first line treatment for MDBO in palliative patients, showing similar clinical and technical success and adverse events (AEs) rate between both techniques. Data about the benefit of this techique in potentially surgical patients is still limited.

Recent retrospective study (Janet J et al, Ann Surg Oncol 2023) and two recent meta-analysis (Barbosa E et al, GIE 2024; Gopakumar H et al, AM J Gastr 2024; both with > 500 cases) found that EUS-CDS group had significantly less technical failure rate and less postprocedure pancreatitis rate.

Thus, our hypothesis is that EUS-CDS has benefits in terms of decreasing those rates (technical failure, postprocedure pancreatitis) when compared to ERCP in MDBO in potentially surgical patients with resectable and borderline disease.

ELIGIBILITY:
Inclusion Criteria:

* Malignant distal biliary obstruction diagnosed in patient considered RESECTABLE or POTENTIALLY RESECTABLE/BORDERLINE with biliary drainage indication: i) impaired hepatic enzymes (including hyperbilirubinemia) x3 times upper the superior normal value. ii) Radiologic singns of extrahepatic bile duct obstruction with presence of retrograde dilatation, of at least 12-mm axial diameter.
* Consensual malignancy by a bilio-pancreatic multidisciplinar committe (histological confirmation is not mandatory)
* Patient capable of understanding and/or singning the informed consent.
* Patient who understands the type of study and will comply with all follow-up tests throughout its duration

Exclusion Criteria:

* Pregnancy or lactation.
* Severe coagulation disorder: INR > 1.5 non correctable with plasma administration and/or platelet count < 50.000/mm3.
* Distal malignant biliary strictures in patients considered directly resectable, non-surgical, unresectable, or palliative
* Benign or uncertain etiology of biliary strictures or strictures located proximally or in close proximity to the hilum.
* Patients with prior biliary stents or other biliary drainages (e.g., PTCD).
* Altered intestinal anatomy due to prior surgery that prevents or hinders papillary access (e.g., gastric bypass, Billroth II, duodenal switch, Roux-en-Y).
* Stenosis in the antral or duodenal region that prevents access to the duodenum and reaching the papilla.
* Situations that do not allow for upper gastrointestinal endoscopy (e.g., esophageal stricture).
* Patients with functional diversity, who lack the capacity to understand the nature and potential consequences of the study, except when a legal representative is available.
* Patients incapable of maintaining follow-up appointments (lack of adherence).
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-06-06 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
Postprocedure surgical challenges rate | 1 day to 24 months
  Percentage of biliary drainage technical failure and/or percentage of postprocedure acute pancreatitis.

SECONDARY OUTCOMES:
Clinical success | 14 days after BD
  In jaundice: decreasing > 50% of bilirrubin or normalization of bilirrubin levels 14 days after endoscopic procedure.
AE - biliary drainage | 0 to 30 days after BD
  Adverse events rate related to biliary drainage according to the AGREE classification
AE - surgery | 0 to 90 days after surgery
  Adverse events rate related to surgery according to the Claiven and Dindo classification.
Delay in days between endoscopic biliary drainage and cephalic duodenopancreatectomy (CDP) | 1 day to 6 months
  Number of days between intervention (T1-biliary drainage) and surgery
Rate of surgery | 1 to 24 months
  Rate of patients that undergo to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joan B Gornals, PhD, Principal Investigator — Hospital Universitari de Bellvitge, SEED
Locations (10):
- Spain (10):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital General Universitario de Castellón, Castellon, Castellón
  - Hospital de Sant Pau i de la Santa Creu, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, Hospitalet de Llobregat, Barcelona, Catalonia
  - Hospital Mútua de Terrassa, Terrassa, Catalonia
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Teoh AYB, Napoleon B, Kunda R, Arcidiacono PG, Kongkam P, Larghi A, Van der Merwe S, Jacques J, Legros R, Thawee RE, Saxena P, Aerts M, Archibugi L, Chan SM, Fumex F, Kaffes AJ, Ma MTW, Messaoudi N, Rizzatti G, Ng KKC, Ng EKW, Chiu PWY. EUS-Guided Choledocho-duodenostomy Using Lumen Apposing Stent Versus ERCP With Covered Metallic Stents in Patients With Unresectable Malignant Distal Biliary Obstruction: A Multicenter Randomized Controlled Trial (DRA-MBO Trial). Gastroenterology. 2023 Aug;165(2):473-482.e2. doi: 10.1053/j.gastro.2023.04.016. Epub 2023 Apr 28. PMID 37121331
- [Background] Janet J, Albouys J, Napoleon B, Jacques J, Mathonnet M, Magne J, Fontaine M, de Ponthaud C, Durand Fontanier S, Bardet SSM, Bourdariat R, Sulpice L, Lesurtel M, Legros R, Truant S, Robin F, Prat F, Palazzo M, Schwarz L, Buc E, Sauvanet A, Gaujoux S, Taibi A. Pancreatoduodenectomy Following Preoperative Biliary Drainage Using Endoscopic Ultrasound-Guided Choledochoduodenostomy Versus a Transpapillary Stent: A Multicenter Comparative Cohort Study of the ACHBT-FRENCH-SFED Intergroup. Ann Surg Oncol. 2023 Aug;30(8):5036-5046. doi: 10.1245/s10434-023-13466-8. Epub 2023 Apr 17. PMID 37069476
- [Background] Chen YI, Sahai A, Donatelli G, Lam E, Forbes N, Mosko J, Paquin SC, Donnellan F, Chatterjee A, Telford J, Miller C, Desilets E, Sandha G, Kenshil S, Mohamed R, May G, Gan I, Barkun J, Calo N, Nawawi A, Friedman G, Cohen A, Maniere T, Chaudhury P, Metrakos P, Zogopoulos G, Bessissow A, Khalil JA, Baffis V, Waschke K, Parent J, Soulellis C, Khashab M, Kunda R, Geraci O, Martel M, Schwartzman K, Fiore JF Jr, Rahme E, Barkun A. Endoscopic Ultrasound-Guided Biliary Drainage of First Intent With a Lumen-Apposing Metal Stent vs Endoscopic Retrograde Cholangiopancreatography in Malignant Distal Biliary Obstruction: A Multicenter Randomized Controlled Study (ELEMENT Trial). Gastroenterology. 2023 Nov;165(5):1249-1261.e5. doi: 10.1053/j.gastro.2023.07.024. Epub 2023 Aug 6. PMID 37549753
- [Background] Barbosa EC, Santo PADE, Baraldo S, Nau AL, Meine GC. EUS- versus ERCP-guided biliary drainage for malignant biliary obstruction: a systematic review and meta-analysis of randomized controlled trials. Gastrointest Endosc. 2024 Sep;100(3):395-405.e8. doi: 10.1016/j.gie.2024.04.019. Epub 2024 Apr 20. PMID 38648989
- [Background] Gopakumar H, Singh RR, Revanur V, Kandula R, Puli SR. Endoscopic Ultrasound-Guided vs Endoscopic Retrograde Cholangiopancreatography-Guided Biliary Drainage as Primary Approach to Malignant Distal Biliary Obstruction: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Am J Gastroenterol. 2024 Aug 1;119(8):1607-1615. doi: 10.14309/ajg.0000000000002736. Epub 2024 Feb 29. PMID 38421018